CLINICAL TRIAL: NCT00003090
Title: Phase II Trial of Bolus Interleukin-2 in Previously Treated Lung Cancer
Brief Title: Biological Therapy in Previously Treated Patients With Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Biotherapy Research Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065794; CBRG-9602; NBSG-9602; NCI-V97-1345
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2000-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill non-small cell lung cancer cells.

PURPOSE: Phase II trial to study the effect of biological therapy with interleukin-2 in patients with previously treated non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and median duration of response of interleukin-2 (IL-2) in patients with previously treated non-small cell lung cancer. II. Determine the median survival of patients treated with IL-2. III. Further delineate the toxicity of IL-2 in these patients.

OUTLINE: This is an open label study. Patients receive bolus interleukin-2 on days 1-5 and 8-12. The cycle repeats every 3 weeks. Patient response is evaluated after 2 cycles. Patients with stable disease, partial, or complete response may be treated with maintenance IL-2 for up to 4 additional cycles. Patient evaluation is performed after every 2 cycles. At this point, patients with stable or responding disease may be treated with IL-2 every 6 weeks until disease progression, intolerable toxic effects, or 2 cycles beyond complete response.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory non-small cell lung cancer At least one prior systemic therapy OR prior radiation therapy Must have measurable disease Previously irradiated sites of disease are not considered evaluable unless there is radiologic documentation of progression

PATIENT CHARACTERISTICS: Age: Not specified Performance Status: ECOG 0-2 Life Expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Hemoglobin greater than 10 g/dL Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 2.0 mg/dL Cardiovascular: No prior history of myocardial infarction within previous 6 months No uncompensated congestive heart failure No primary (not due to electrolytes or drugs) cardiac arrhythmias besides premature ventricular contractions Pulmonary: No dyspnea at rest or need for supplemental oxygen Patients with symptomatic lung disease or extensive lung metastases must have oxygen saturation greater than 90% Other: Not pregnant or nursing Negative pregnancy test Patients with elevated temperatures greater than 100.5 F must have no occult infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent cyclosporin Chemotherapy: At least 3 weeks since chemotherapy and recovered No concurrent methotrexate See Disease Characteristics Endocrine therapy: No concurrent systemic corticosteroids Radiotherapy: At least 3 weeks since radiotherapy See Disease Characteristics Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: Datchen F. Tai, MD, Study Chair — Cancer Biotherapy Research Group
Locations (3):
- United States (3):
  - Bloomington Hospital, Bloomington, Indiana
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - St. Joseph Regional Cancer Center, Bryan, Texas